CLINICAL TRIAL: NCT01623141
Title: Correlation Between 3 Phase Bone Scintigraphy and Pressure Pain Thresholds in Patients With CRPS
Brief Title: Correlation Between 3 Phase Bone Scintigraphy and Pressure Pain Thresholds in Patients With Complex Regional Pain Syndrome (CRPS)
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Christoph Maier, Prof. Dr. med. (Head of the pain clinic of the Bergmannsheil University Hospital), Ruhr University of Bochum
Other Study IDs: Scinti/PressurePain2011
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Complex Regional Pain Syndrome Type I of the Upper Limb; Unilateral Limb Pain of Other Origin; Healthy Subjects
Keywords: CRPS; TPBS; Pressure pain thresholds; limb pain of other origin
MeSH Terms: conditions — Reflex Sympathetic Dystrophy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with CRPS: 18 patients with unilateral CPRS of the upper limb were included to the study
  Interventions: Procedure: Pressure Pain measurement
- Patients with limb pain of other origin: 17 patients with unilateral upper limb pain of other origin served as control group
  Interventions: Procedure: Pressure Pain measurement
- Healthy subjects: 18 healthy subjects were included to establish reference data for the pressure pain thresholds
  Interventions: Procedure: Pressure Pain measurement

INTERVENTIONS:
Procedure: Pressure Pain measurement — The pressure pain thresholds were established using a manual pressure algometer. The investigated joints were the carpus, the metacarpophalangeal and the proximal interphalangeal joints
  Other Names: SOMEDIC Production AB, Sweden, Algometer Type II

SUMMARY:
The aim of the study is to investigate the correlation between increased bone metabolism in the 3 phase bone scintigraphy (TPBS) and decreased pressure pain thresholds in patients with complex regional pain syndrome (CRPS) of the upper limb and a non-CRPS-group. The investigators assume that there will be a significant correlation between the investigated values in the CRPS-group whereas the non-CRPS-group shows no significant correlation.

DETAILED DESCRIPTION:
Pressure pain of the distal hand joints is a predominant symptom of CRPS. But so far, the diagnostic value of pressure pain in the diagnosis of CRPS has not been investigated. We compared the pressure pain thresholds of the carpus, metacarpophalangeal and proximal interphalangeal joints to a region of interest-based (ROI) analysis of a TBPS in patients with CRPS and patients with limb pain of other origin (non-CRPS-group).Additionally, the PPTs were established for a healthy control group to get reference data.

ELIGIBILITY:
Inclusion Criteria:

every participant:

* aged > 18 years with written informed consent
* adequate understanding of the german language
* indication for a TPBS independent of the study

Patients with CRPS:

* patients with CRPS type 1 of the upper limb diagnosed on the basis of the budapest criteria (Harden, Bruehl et al., 2010)
* unilateral pain

Control group:

* patients with pain of the upper limbs of other origin than CRPS who underwent a TPBS
* unilateral pain

Healthy subjects:

* checked by the DFNS IMI questionnaire

Exclusion Criteria:

* missing informed consent
* inadequate understanding of the german language
* disease duration of more than 12 months
* other disease of the upper extremity (e.g. polyarthrosis, rheumatoid arthritis)
* pregnancy/ lactation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study sample consists of three groups:
  1. Patients with CRPS of one of the upper limb type 1 (n=18)
  2. Patients with unilateral upper limb pain of other origin (n=17)
  3. Healthy subjects (n=18)
  All patients were recruited from the Department of Pain medicine and the Department of nuclear medicine of the University Hospital Bergmannsheil
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Decrease of the pressure pain thresholds of the distal hand joints | half an hour
  The pressure pain thresholds (PPT) were mesured for the carpus, metacarpophalangeal and proximal interphalangeal joints of both hands. The mean of three determined measurements of each joint was taken as the final value. Subseqently the PPT were compared to the results of the 3 phase bone scintigraphy and the reference data of the healthy subjects.

SECONDARY OUTCOMES:
Increased bone metabolism in the 3 phase bone scintigraphy | 3 hours
  All Patients with CRPS and limb pain of other origin underwented a 3 phase bone scitigraphy to investigate a possible increased bone metabolism. Phase one and two were recorded within the first five minutes after injection of approximately 500-700 MBq 99mTechnetium-labeled methylene diphosphonate. The third phase was obtained two to three hours after injection.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Maier, Prof. Dr., Study Director — Head of the pain clinic of the Bergmannsheil University Hospital
Locations (1):
- Bergmannsheil, department for pain management, Bochum, North Rhine-Westphalia, Germany